CLINICAL TRIAL: NCT02045004
Title: Association Between Changes in Cerebral Gray Matter Volume and Postoperative Cognitive Dysfunction in Elderly Patients Following Sevoflurane Anesthesia (POCD-MRI)
Brief Title: Cohort Study to Investigate the Association Between Changes in Brain Volume and Postoperative Cognitive Dysfunction
Acronym: POCD-MRI
Status: Completed | Type: Observational
Sponsor: Nicolai Goettel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Nicolai Goettel, MD, Staff Anesthesiologist, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: POCD-MRI
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Cognitive Dysfunction; Delirium; Dementia
Keywords: Anesthesia; Surgery; Geriatrics; Postoperative cognitive dysfunction; Postoperative delirium; Dementia; Postoperative complications; Neurological complications; Psychological complications
MeSH Terms: conditions — Postoperative Cognitive Complications; Delirium; Dementia; Emergence Delirium; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery Group Sevoflurane: Patients aged ≥ 65 years undergoing major surgical procedures.
- Control Group: Healthy study participants aged ≥ 65 years (no surgical intervention).

SUMMARY:
Despite an ongoing controversy in the scientific literature, the link between anesthesia and dementia and/or cerebral atrophy remains unclear. Recent retrospective data suggests an association of surgery with a reduction in brain volume. With the present prospective cohort study, we would like to reproduce and verify these results, and investigate a possible association with the postoperative cognitive performance.

We will measure cerebral gray matter volumes in elderly patients before, 3 and 12 months after major non-cardiac surgery and determine cognitive functions at the same time.

Study hypothesis:

1. Surgery under general anesthesia in elderly patients is associated with a loss of gray matter.
2. The degree of cognitive dysfunction is associated with the loss of grey matter in brain areas relevant for cognitive functions.

DETAILED DESCRIPTION:
Background:

Anesthesia care for elective surgery of patients that are in their seventies or eighties is an ever-growing entity in clinical practice, given the demographic development in many countries of the Western world. Cognitive decline of variable degree is frequently observed after major surgery in elderly patients. A potential association between anesthesia and the development of dementia and brain atrophy in elderly patients is controversial. However, it is not uncommon that during preoperative visits by the anesthesiologist, patients express fear to suffer some sort of cognitive decline after the operation, and raise concerns about psychological or neurological long-term adverse effects (e.g. memory loss) related to anesthesia. Clinicians have identified this problem decades ago, and are adding postoperative cognitive dysfunction (POCD) to the list of frequent complications of anesthesia in elderly patients; yet, there is a lack of prospective clinical data and poor understanding of the pathophysiology of POCD, and no preventive strategy or treatment has been described so far.

One study reported an incidence of postoperative cognitive dysfunction (POCD) of 41% in surgical patients 60 years of age, or older. In a previous study conducted by our group, as many as 47% of patients over 65 years presented with POCD one week after surgery. In many patients, this is a transient problem, but some patients retain permanent deficits, with increased mortality and important consequences on the socioeconomic situation. An association between surgery and long-term cognitive decline has not been established yet; however, patients who develop postoperative delirium (a transient, but particularly severe form of POCD) have an increased risk of developing dementia in the years following surgery. However, in a cohort follow-up study, the diagnosis of POCD itself did not represent a significant risk factor for dementia. The pathophysiology of postoperative cognitive decline remains unclear. However, studies in animals have shown that the systemic inflammatory response elicited by the surgical procedure is associated with microglial activation and postoperative cognitive impairment. Furthermore, volatile anesthetics have been shown to be neurotoxic in cell cultures, and in some animal experiments exposure to clinical concentrations of volatile anesthetics was associated with postoperative cognitive decline. A recent retrospective analysis of cohort data suggests that surgery may be associated with a decrease in brain volume in patients. However, due to methodological limitations in this study, no analysis of a potential link between atrophy and cognitive functions was made.

Study Design:

Prospective cohort study

Study Groups:

Two groups of patients will be investigated. Seventy patients undergoing major surgical procedures will be recruited for this study, and 30 healthy study participants (no surgical intervention) will be recruited to serve as controls. In all patients, baseline cognitive functions and structural MRI imaging including determination of gray matter volumes relevant for cognitive functions (hippocampus) will be performed.

* Group 1: Surgery group Sevoflurane (n = 70)
* Group 2: Control group (n = 30)

Recruitment:

Study participants of the Surgery group Sevoflurane (Group 1) will be recruited as patients of the Basel University Hospital, a tertiary medical care center in Basel, Switzerland, associated with the University of Basel, Switzerland. Study participants of the Control group (Group 2) will be recruited randomly.

Endpoints:

Targeted primary endpoint of the study is the difference in change of hippocampal volume over time between patients with POCD and patients without POCD.

Secondary endpoint is the correlation between change in cerebral volume and change in cognitive function.

Anesthetic Management:

Anesthesia will be standardized (general anesthesia using sevoflurane and fentanyl for maintenance, thiopental for induction and atracurium or rocuronium for neuromuscular blockade). Intraoperatively, the dose of anesthetics will be controlled using an EEG derived index (depth of anesthesia monitoring (Bispectral Index (BIS), Aspect Medical Systems), and end-tidal sevoflurane concentration monitoring). Furthermore, intraoperative bilateral cerebral near-infrared spectroscopy (NIRS) monitoring (NIRO-200, Hamamatsu Photonics, Japan) will be applied. Data will be downloaded directly from the monitors and the anesthesia machine (Dräger Perseus) using ICM+ software.

Neuropsychological Assessment:

The cognitive assessment test battery CERAD-Plus consistent of the Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB), Trail Making Tests A+B, and phonetic fluency (s-words), as well as the Test for Attentional Performance (TAP) developed to analyze different aspects of attention, will be performed preoperatively, at 7 days, 3 month and 12 months postoperatively. Training of all study personnel and supervision of cognitive testing will be carried out by the Memory Clinic at Basel University Hospital. Cognitive functions will be quantified using the CERAD total score, in its demographically corrected form. A correction for short-term practice effects will be carried out based on previous work.

Blood Samples:

Blood samples will be taken from study participants preoperatively, 12h postoperatively, and on day 2 and 7, to determine levels of C-reactive protein (CRP), interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-alpha). Blood samples will be stored for 1 year to allow additional determinations.

Demographic, Procedural and Subjective Patient Data:

* Age, sex, and years of education.
* Cognitive testing as outlined: CERAD-Plus (CERAD-NAB, Trail Making Tests A+B, phonetic fluency (s-words)), Test for Attentional Performance (TAP), preoperatively, at 7 days, 3 months and 12 months postoperatively.
* Charlson Comorbidity Score preoperatively, at 3 months and 1 year postoperatively
* Instrumental Activities of Daily Living (IADL) preoperatively, at 3 months and 1 year postoperatively.
* Geriatric Depression Scale (GDS) preoperatively, at 3 months and 1 year postoperatively.
* Short Form Health Survey (SF-36) preoperatively, at 3 months and 1 year postoperatively.
* ASA physical status, type and duration of anesthesia, type and duration of surgery.
* Postoperative delirium (Confusion Assessment Method; CAM), repeat surgery and postoperative infections.
* Subjective grading of cognitive functions on a VAS scale (0-10) preoperatively, at 7 days, 3 months and 1 year postoperatively.
* Subjective grading of change in cognitive functions on a five-point Likert scale (much worse, worse, equal, better, much better) at 7 days, 3 months and 1 year postoperatively.
* Subjective grading of successful surgery (Yes/No) at 7 days, 3 months and 1 year postoperatively.
* Subjective grading of pain on a VAS scale (0-10) preoperatively, 7 days, 3 months and 1 year postoperatively.

Magnetic Resonance Imaging (MRI):

MRI will be performed preoperatively, at 3 months, and 1 year postoperatively on the same day as cognitive function testing. No intravenous contrast dye will be administered. Training of all study personnel and MRI evaluation, and/or supervision of MRI evaluation, will be carried out by the Division of Neuroradiology at the University Hospital Basel. High resolution anatomic and diffusion MRI will be performed using the hospital's 3T MAGNETOM Prisma™ MRI scanner (Siemens, Zurich, Switzerland). For our initial MRI analysis, we assume that the same regions as those described in mild cognitive impairment (MCI) and Alzheimer's disease (AD) are relevant to POCD. We will perform a region of interest (ROI) analysis during this part of the analysis. In a second step, we will perform a whole brain analysis.

The whole brain MRI protocol includes high resolution three-dimensional (3D)-T1 (MPRAGE sequence, repetition time (TR) = 1620 ms, echo time (TE) = 2.48 ms, 192 slices), clinical standard at the University Hospital Basel) and 3D-T2 (SPACE sequence, TR = 3200 ms, TE = 408 ms, 192 slices) imaging for segmentation. Furthermore, a diffusion sequence (DTI sequence, TR = 5800 ms, TE = 77 ms, 50 slices, 64 directions, 8 B0) for quantitative imaging will be used. We added a two-dimensional (2D)-PD/T2 weighted sequence (TSE sequence, TR = 4480 ms, TE1 = 9 ms, TE2 = 106 ms, 46 slices) for diagnostic purposes. The total acquisition time for the MRI is approximately 24 minutes.

Statistical Analysis:

Cortical reconstruction and volumetric segmentation will be performed with the FreeSurfer image analysis suite, which is documented and freely available for download online (http://surfer.nmr.mgh.harvard.edu/). The technical details of these procedures are described in prior publications.

Comparisons (preoperatively to 3 months postoperatively) of hippocampal volume and the results of voxel-based volumetry of the medio-temporal lobe and lateral association areas of the temporal and parietal lobes will be performed using region of interest (ROI) analysis. The quantitative imaging results will be correlated to the CERAD total score performance obtained on the same day as the MRI scans. The relationship of changes in volume (if present) with intraoperative depth of anesthesia (BIS) and the administered dose of sevoflurane expressed as age-corrected minimum alveolar concentration (MAC) equivalent multiplied by time of administration will be calculated. We will also use multivariate approaches (voxel-wise multivariate analysis (MANOVA) and classification/prediction procedure) on multi-parameter MRI data in order to build optimal composite predictors of patients' neuropsychological outcomes. In whole brain analysis, we will use a multiple regression and repeated measures ANOVA whole brain voxel-wise analyses in FreeSurfer to correlate the estimated modulated gray matter volume with the neuropsychological scores.

Sample Size Calculation:

Assuming that 41% of operated patients develop POCD, and a standard deviation of the hippocampal volume change of 0.45 in both patients with POCD and without POCD, a total sample size of 56 subjects may detect a difference of 0.4 mm3 in hippocampal volume with a power of 90% at a two-sided significance level of 5%. To compensate for the high loss to follow-up which is unfortunately typical for studies on POCD, and estimated at 20%, we will recruit 70 patients in the surgery group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Elective major surgery
* Planned general anesthesia

Exclusion Criteria:

* Cardiac surgery
* Neurosurgery including carotid endarterectomy
* Preoperative Mini Mental State (MMS) Examination Score < 24
* Previous pathological neuroimaging (if available)
* History of cerebral or cerebrovascular pathology
* Chronic use of psychiatric medication
* Alcohol or substance abuse
* A history of chronic pain unrelated to the planned surgery
* Any contraindication for MRI (e.g. pacemakers and other MR-incompatible metal implants)
* Claustrophobia
* Lack of informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Study participants in Group 1 (Surgery group Sevoflurane) will be recruited as patients of the Basel University Hospital, a tertiary medical center affilitated to the University of Basel, Switzerland. Study participants in Group 2 (Control group) will be recruited randomly from the local population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Cerebral gray matter volume | Preoperatively, at 3 month and 12 month postoperatively
  Hippocampal volume is specifically assessed.

SECONDARY OUTCOMES:
Cognitive function | Preoperatively, at 7 days, 3 month and 12 month postoperatively
  The neuropsychological assessment test battery CERAD-Plus consistent of the Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB), Trail Making Tests A+B, and phonetic fluency (s-words), as well as the Test for Attentional Performance (TAP) developed to analyze different aspects of attention, will be performed. Cognitive functions will be quantified using the CERAD total score, in its demographically corrected form.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — Department of Anesthesia, University Hospital Basel, Switzerland; Luzius A Steiner, MD, PhD, Study Chair — Department of Anesthesia, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burkhart CS, Steiner LA. Can postoperative cognitive dysfunction be avoided? Hosp Pract (1995). 2012 Feb;40(1):214-23. doi: 10.3810/hp.2012.02.962. PMID 22406897
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Avidan MS, Searleman AC, Storandt M, Barnett K, Vannucci A, Saager L, Xiong C, Grant EA, Kaiser D, Morris JC, Evers AS. Long-term cognitive decline in older subjects was not attributable to noncardiac surgery or major illness. Anesthesiology. 2009 Nov;111(5):964-70. doi: 10.1097/ALN.0b013e3181bc9719. PMID 19786858
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Steinmetz J, Siersma V, Kessing LV, Rasmussen LS; ISPOCD Group. Is postoperative cognitive dysfunction a risk factor for dementia? A cohort follow-up study. Br J Anaesth. 2013 Jun;110 Suppl 1:i92-7. doi: 10.1093/bja/aes466. Epub 2012 Dec 28. PMID 23274780
- [Background] Terrando N, Monaco C, Ma D, Foxwell BM, Feldmann M, Maze M. Tumor necrosis factor-alpha triggers a cytokine cascade yielding postoperative cognitive decline. Proc Natl Acad Sci U S A. 2010 Nov 23;107(47):20518-22. doi: 10.1073/pnas.1014557107. Epub 2010 Nov 1. PMID 21041647
- [Background] Wan Y, Xu J, Ma D, Zeng Y, Cibelli M, Maze M. Postoperative impairment of cognitive function in rats: a possible role for cytokine-mediated inflammation in the hippocampus. Anesthesiology. 2007 Mar;106(3):436-43. doi: 10.1097/00000542-200703000-00007. PMID 17325501
- [Background] Cerejeira J, Firmino H, Vaz-Serra A, Mukaetova-Ladinska EB. The neuroinflammatory hypothesis of delirium. Acta Neuropathol. 2010 Jun;119(6):737-54. doi: 10.1007/s00401-010-0674-1. Epub 2010 Mar 24. PMID 20309566
- [Background] van Gool WA, van de Beek D, Eikelenboom P. Systemic infection and delirium: when cytokines and acetylcholine collide. Lancet. 2010 Feb 27;375(9716):773-5. doi: 10.1016/S0140-6736(09)61158-2. PMID 20189029
- [Background] Eckenhoff RG, Johansson JS, Wei H, Carnini A, Kang B, Wei W, Pidikiti R, Keller JM, Eckenhoff MF. Inhaled anesthetic enhancement of amyloid-beta oligomerization and cytotoxicity. Anesthesiology. 2004 Sep;101(3):703-9. doi: 10.1097/00000542-200409000-00019. PMID 15329595
- [Background] Culley DJ, Baxter MG, Crosby CA, Yukhananov R, Crosby G. Impaired acquisition of spatial memory 2 weeks after isoflurane and isoflurane-nitrous oxide anesthesia in aged rats. Anesth Analg. 2004 Nov;99(5):1393-1397. doi: 10.1213/01.ANE.0000135408.14319.CC. PMID 15502036
- [Background] Kline RP, Pirraglia E, Cheng H, De Santi S, Li Y, Haile M, de Leon MJ, Bekker A; Alzheimer's Disease Neuroimaging Initiative. Surgery and brain atrophy in cognitively normal elderly subjects and subjects diagnosed with mild cognitive impairment. Anesthesiology. 2012 Mar;116(3):603-12. doi: 10.1097/ALN.0b013e318246ec0b. PMID 22293721
- [Background] Baranov D, Bickler PE, Crosby GJ, Culley DJ, Eckenhoff MF, Eckenhoff RG, Hogan KJ, Jevtovic-Todorovic V, Palotas A, Perouansky M, Planel E, Silverstein JH, Wei H, Whittington RA, Xie Z, Zuo Z; First International Workshop on Anesthetics and Alzheimer's Disease. Consensus statement: First International Workshop on Anesthetics and Alzheimer's disease. Anesth Analg. 2009 May;108(5):1627-30. doi: 10.1213/ane.0b013e318199dc72. PMID 19372347
- [Background] Seitz DP, Shah PS, Herrmann N, Beyene J, Siddiqui N. Exposure to general anesthesia and risk of Alzheimer's disease: a systematic review and meta-analysis. BMC Geriatr. 2011 Dec 14;11:83. doi: 10.1186/1471-2318-11-83. PMID 22168260
- [Background] Smielewski P, Czosnyka M, Steiner L, Belestri M, Piechnik S, Pickard JD. ICM+: software for on-line analysis of bedside monitoring data after severe head trauma. Acta Neurochir Suppl. 2005;95:43-9. doi: 10.1007/3-211-32318-x_10. PMID 16463818
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064
- [Background] Chandler MJ, Lacritz LH, Hynan LS, Barnard HD, Allen G, Deschner M, Weiner MF, Cullum CM. A total score for the CERAD neuropsychological battery. Neurology. 2005 Jul 12;65(1):102-6. doi: 10.1212/01.wnl.0000167607.63000.38. PMID 16009893
- [Background] Ehrensperger MM, Berres M, Taylor KI, Monsch AU. Early detection of Alzheimer's disease with a total score of the German CERAD. J Int Neuropsychol Soc. 2010 Sep;16(5):910-20. doi: 10.1017/S1355617710000822. Epub 2010 Aug 4. PMID 20682088
- [Background] Burkhart CS, Birkner-Binder D, Gagneux A, Berres M, Strebel SP, Monsch AU, Steiner LA. Evaluation of a summary score of cognitive performance for use in trials in perioperative and critical care. Dement Geriatr Cogn Disord. 2011;31(6):451-9. doi: 10.1159/000329442. Epub 2011 Jul 20. PMID 21778726
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] McHorney CA. Measuring and monitoring general health status in elderly persons: practical and methodological issues in using the SF-36 Health Survey. Gerontologist. 1996 Oct;36(5):571-83. doi: 10.1093/geront/36.5.571. PMID 8942101
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Helms G, Draganski B, Frackowiak R, Ashburner J, Weiskopf N. Improved segmentation of deep brain grey matter structures using magnetization transfer (MT) parameter maps. Neuroimage. 2009 Aug 1;47(1):194-8. doi: 10.1016/j.neuroimage.2009.03.053. Epub 2009 Mar 31. PMID 19344771
- [Background] Kherif F, Poline JB, Flandin G, Benali H, Simon O, Dehaene S, Worsley KJ. Multivariate model specification for fMRI data. Neuroimage. 2002 Aug;16(4):1068-83. doi: 10.1006/nimg.2002.1094. PMID 12202094
- [Background] Mapleson WW. Effect of age on MAC in humans: a meta-analysis. Br J Anaesth. 1996 Feb;76(2):179-85. doi: 10.1093/bja/76.2.179. PMID 8777094
- [Background] Liu Y, Paajanen T, Zhang Y, Westman E, Wahlund LO, Simmons A, Tunnard C, Sobow T, Mecocci P, Tsolaki M, Vellas B, Muehlboeck S, Evans A, Spenger C, Lovestone S, Soininen H; AddNeuroMed Consortium. Combination analysis of neuropsychological tests and structural MRI measures in differentiating AD, MCI and control groups--the AddNeuroMed study. Neurobiol Aging. 2011 Jul;32(7):1198-206. doi: 10.1016/j.neurobiolaging.2009.07.008. Epub 2009 Aug 14. PMID 19683363
- [Background] Rasmussen LS, Larsen K, Houx P, Skovgaard LT, Hanning CD, Moller JT; ISPOCD group. The International Study of Postoperative Cognitive Dysfunction. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89. doi: 10.1034/j.1399-6576.2001.045003275.x. PMID 11207462
- [Derived] Goettel N, Mistridis P, Berres M, Reinhardt J, Stippich C, Monsch AU, Steiner LA. Association between changes in cerebral grey matter volume and postoperative cognitive dysfunction in elderly patients: study protocol for a prospective observational cohort study. BMC Anesthesiol. 2016 Nov 25;16(1):118. doi: 10.1186/s12871-016-0285-z. PMID 27884107